CLINICAL TRIAL: NCT06016660
Title: Acute Effect of Resistance Exercise, Neuromuscular Electrical Stimulation, and Transcutaneous Electrical Stimulation Applications on Muscle Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Barış SEVEN, Ph.D. research assistant, Gazi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EMGHealthy
Record Dates: First submitted 2023-06-07; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resistance exercise (Experimental): Resistance exercise
  Interventions: Other: Physiotherapy
- Neuromuscular electrical stimulation (Experimental): Neuromuscular electrical stimulation
  Interventions: Other: Physiotherapy
- Transcutaneous electrical stimulation (Experimental): Transcutaneous electrical stimulation
  Interventions: Other: Physiotherapy
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Physiotherapy — Resistance exercise, Neuromuscular electrical stimulation, and Transcutaneous electrical stimulation
  Arms: Neuromuscular electrical stimulation; Resistance exercise; Transcutaneous electrical stimulation

SUMMARY:
The aim of our study is to investigate the effects of single-session resistance exercise, neuromuscular electrical stimulation, and transcutaneous electrical stimulation on the level of muscle activation and their superiority over each other on both the ipsilateral and contralateral sides. Our randomized controlled crossover study included 21 participants (13 female, 8 male, age; 27.7±4). Transcutaneous electrical stimulation was used for sensory input. A single-session application was performed only to the right extremities of all participants, and the acute effects on muscle activation on both the ipsilateral and contralateral sides were evaluated. Muscle activation was evaluated with superficial EMG. SPSS® Statistics V22.0 software was used for statistical analysis. As a result of the statistical analysis, a significant increase in activation was found only in the sensory input application group on the ipsilateral side flexor carpi radialis (FCR) (p=0.001), flexor carpi ulnaris (FCU) (p<0.001), flexor digitorum superficialis (FDS) (p=0.023) and flexor digitorum profundus (FDP) (p=0.003) muscles. On the contralateral side, there was an increase in activation in all muscles (FCR; p<0.001, FCU; p=0.033, FDS; p=0.017 and FDP; p=0.001) in the resistant exercise group. In addition, there was a significant increase in the activation of certain muscles on the contralateral side in the NMES application group (FCR (p=0.049) and FDP (p=0.016) muscles) and the sensory input application group (FDP (p=0.004) and FDS (p=0.043) muscles). In situations where movement is contraindicated, ipsilateral sensory input can increase the level of muscle activation through both cortical and peripheral neural mechanisms.In addition, resistance exercise to be performed on the contralateral side can be an effective application to increase muscle activation on the ipsilateral side.

ELIGIBILITY:
Inclusion Criteria:

• After providing detailed information about the study, individuals who had agreed to participate in the research were included in the study.

Exclusion Criteria:

* Individuals with any central or peripheral nervous system disease/injury affecting the upper extremity,
* Individuals with a history of orthopedic injury that could impact the study,
* Individuals with a history of neuromuscular disease, congenital anomalies, skin infections, or cognitive impairments,
* Individuals with a history of systemic or metabolic diseases that could potentially affect the study,
* Individuals with a body mass index (BMI) above 30 kg/m2.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Superficial electromyography | through study completion, an average of 1 year
  Muscle activation measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Barış SEVEN, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No